CLINICAL TRIAL: NCT04270617
Title: A Prospective, Randomized-controlled Study to Evaluate the Effect of a Standardized Yoga Practice on Chronic Back Pain
Brief Title: The Effect of Yoga Practice on Chronic Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-00824
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): The control arm will involve usual care - 6 weeks of physical therapy, NSAIDs, and epidural steroid injections
- Yoga Arm (Experimental): The study arm will involve a yoga protocol devised by Eddie Stern - a renowned Ashtanga yoga practitioner, and can include NSAIDs.
  Interventions: Behavioral: Yoga program

INTERVENTIONS:
Behavioral: Yoga program — The intervention will be a 6-week ashtanga yoga program designed by world-renowned yogi Eddie Stern. Eddie Stern is an internationally known Ashtanga yoga teacher, in independent practice not affiliated with NYULH, who has done significant work exploring the physiology and science of yoga. He is not currently engaged in his own research. The yoga protocol for chronic back pain was designed with poses specific to addressing core strength but are gentle enough for patients in pain. The protocol is designed to be directed by a teacher initially but can be done at home and is only 18 minutes in duration.
  Arms: Yoga Arm

SUMMARY:
Chronic low back pain is notoriously difficult to treat and is a primary contributor to lost work days and excessive health expenditures, and whose treatment has, in part, contributed to the opioid crisis. Surgery is only an option in a minority of these patients, usually confined to those with structural instability. Yoga is an ancient modality whose benefits are currently being studied.

DETAILED DESCRIPTION:
The purpose of this research study is to determine whether a 6 week standardized yoga practice is superior to usual conservative therapies in the treatment of chronic back pain at 6 months. There is enough data that the most recent ACP guidelines have included yoga as a treatment for chronic back pain, but more data needs to be generated regarding the efficacy of this modality in treating the chronic back pain population.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to and ability to participate in study procedures
* Chronic back pain (pain above the gluteal cleft of at least 3 months duration)

Exclusion Criteria:

* Indication for surgery (i.e., fracture, infection, scoliosis, spondylolisthesis)
* Cardiac, pulmonary or other medical comorbidities that preclude participation in yoga practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in VAS(visual analog scale) | Enrollment visit, 6 months after enrollment visit
  The visual analogue scale or visual analog scale (VAS) is designed to measure pain intensity with less pain being experienced by those in the intervention group in comparison to the control group.
Changes in ODI (Oswestry Disability Index) | Enrollment visit, 6 months after enrollment visit
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. Improvement will be measured by the lower score out of a 100, which reflects less disability.
Changes in SF-36 (Short Form (36) Health Survey ) | Enrollment visit, 6 months after enrollment visit
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. Improvement with those with Yoga will be seen by higher scores in SF-36 which indicate lower disability.

SECONDARY OUTCOMES:
Long term changes in VAS after intervention | Baseline Visit, 6 weeks Visit , 3 months Visit , 1 year Visit , 2 years Visit
  The visual analogue scale or visual analog scale (VAS) is designed to measure pain intensity with less pain being experienced by those in the intervention group in comparison to the control group.
Long term changes in ODI after intervention | Baseline Visit, 6 weeks Visit , 3 months Visit , 1 year Visit , 2 years Visit
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. Improvement will be measured by the lower score out of a 100, which reflects less disability.
Long term changes in SF-36 after intervention | Baseline Visit, 6 weeks Visit , 3 months Visit , 1 year Visit , 2 years Visit
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. Improvement with those with Yoga will be seen by higher scores in SF-36 which indicate lower disability.

CONTACTS AND LOCATIONS:
Overall Officials: Erich Anderer, Principal Investigator — NYU Langone Health
Locations (1):
- NYULangone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to jadie.detolla@nyulangone.org To gain access, data requestors will need to sign a data access agreement.